CLINICAL TRIAL: NCT05795296
Title: Clinical Study of Fruquintinib in Combination With Sintilimab as a First-line Therapy in Gastric Adenocarcinoma/Adenocarcinoma of Esophagogastric Junction
Brief Title: Efficacy and Safety of Fruquintinib With Sintilimab as First-line Therapy in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yingchun Xu, Dr., RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-SH-GC-101
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib+Sintilimab (Experimental): Fruquintinib: 5mg po, d1-d14, q3w
  Sintilimab: 200mg ivgtt, d1, q3w
  Interventions: Drug: Fruquintinib; Drug: Sintilimab

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib: 5mg po, d1-d14, q3w
Drug: Sintilimab — Sintilimab: 200mg ivgtt, d1, q3w

SUMMARY:
The goal of this clinical trial is to explore the efficacy and safety in patients with gastric adenocarcinoma or adenocarcinoma of esophagogastric junction. The main questions it aims to answer are:

* Does this therapy have a promising efficacy?
* Does this therapy have a manageable toxicity? Participants will receive fruquintinib plus sintilimab as first-line therapy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed advanced, recurrent, of metastatic gastric adenocarcinoma or adenocarcinoma of esophagogastric junction;
* ECOG PS: 0-2;
* Adequate hepatic, renal, heart, and hematologic functions;
* At least one measurable lesion (according to RECIST1.1);
* Haven't received any systematic treatment for the cancer involved;
* Expected survival > 12 weeks;
* Contraception until 6 months after the study termination;
* Signed informed consent.

Exclusion Criteria:

* Her-2-positive gastric cancer, or exposed to any immune checkpoint inhibitor;
* Participated in another study;
* Immunodeficiency;
* Received allograft；
* Unmanageable hypertension, diabetes, or coronary disease;
* Have difficulty in taking medicine, or active bleeding;
* Pulmonary tuberculosis, or interstitial lung disease that needs steroid therapy;
* Infection of HIV, HBV, HCV, or other unmanageable infection;
* Other malignant tumor history;
* Allergic to the test drug;
* Other diseases which will affect the results of this study;
* Received resection of stomach;
* Taking anti-tumor traditional Chinese Medicine;
* Severe active bleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months
  The proportion of patients with complete response or partial response, using RECIST v 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 12 months
  Time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Overall survival (OS) | 12 months
  Time from randomization to death from any cause.
Disease Control Rate (DCR) | 12 months
  The proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1.
Adverse Events | 12 months
  Adverse event assessed according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Shuiping Tu, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.